CLINICAL TRIAL: NCT04548596
Title: NOninVasive Intracranial prEssure From Transcranial doppLer Ultrasound Development of a Comprehensive Database of Multimodality Monitoring Signals for Brain-Injured Patients
Acronym: NOVEL ICP
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Collaborators: University of California, San Francisco (Other); National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Responsible Party: Principal Investigator, Xiao Hu, Acting Professor, Emory University
Other Study IDs: STUDY00004039; Pro00105151 (Other: Duke University); R01NS106905 (NIH)
Record Dates: First submitted 2020-09-03; First posted 2020-09-14 (Actual); Last update posted 2025-09-18 (Actual); Status verified 2025-09

CONDITIONS: Traumatic Brain Injury; Subarachnoid Hemorrhage; Intracerebral Hemorrhage; Liver Failure; Ischemic Stroke
MeSH Terms: conditions — Brain Injuries, Traumatic; Subarachnoid Hemorrhage; Cerebral Hemorrhage; Liver Failure; Ischemic Stroke | interventions — Ultrasonography, Doppler, Transcranial

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Transcranial Doppler — In this study, the investigators will primarily use the monitor mode of the Transcranial Doppler (TCD, non-invasive FDA approved device) to record cerebral blood flow velocity (CBFV) signals from the Middle Cerebral Artery and Internal Carotid Artery. TCD data and intracranial pressure (ICP) data will be collected in the following four scenarios. Each recording is up to 60 minutes in length:
  External ventricular drain (EVD) closed to drainage for a 24 hour period as part of the EVD weaning protocol per standard of care (SOC): The Initial reading will be done within 4 hours of EVD closing. The second reading will be done within 4 hours of anticipated removal of EVD.
  EVD closed most of the time and opened to drainage when the ICP becomes elevated per SOC
  EVD with Intra-Parenchymal fiber optical ICP sensor per SOC
  Intra-Parenchymal fiber optical ICP sensor per SOC

SUMMARY:
This is an observational study in neurocritical care units at University of California San Francisco Medical Center (UCSFMC), Zuckerberg San Francisco General Hospital (ZSFGH), UC Davis, and Emory University. In this study, the investigators will primarily use the monitor mode of the Transcranial Doppler (TCD, non-invasive FDA approved device) to record cerebral blood flow velocity (CBFV) signals from the Middle Cerebral Artery and Internal Carotid Artery. TCD data and intracranial pressure (ICP) data will be collected in the following four scenarios. Each recording is up to 60 minutes in length.

Multimodality high-resolution physiological signals will be collected from brain injured patients: traumatic brain injury, subarachnoid and intracerebral hemorrhage, liver failure, and ischemic stroke. This is not a hypothesis-driven study but rather a signal database development project with a goal to collect multimodality brain monitoring data to support development and validation of algorithms that will be useful for future brain monitoring devices. In particular, the collected data will be used to support:

Development and validation of noninvasive intracranial pressure (nICP) algorithms.

Development and validation of continuous monitoring of neurovascular coupling state for brain injury patients

Development and validation of noninvasive approaches of detecting elevated ICP state.

Development and validation of approaches to determine most likely causes of ICP elevation.

Development and validation of approaches to detect acute cerebral hemodynamic response to various neurovascular procedures.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects 18 years of age and older
2. Subjects who have an ICP Monitoring device

Exclusion Criteria:

1. Unstable medical illness such as recordings might interfere with medical care.
2. Subjects that don't have a viable temporal window to insonate the MCA.
3. Subjects that have skull fractures that the attending or study investigators believe participation would add clinical risk to the subject.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The investigators aim to collect multimodality high-resolution physiological signals from brain injured patients: traumatic brain injury, subarachnoid and intracerebral hemorrhage, liver failure, and ischemic stroke.
Sampling Method: Non-Probability Sample
Enrollment: 162 (Actual)
Dates: Start 2014-09-10 (Actual); Primary Completion 2025-04-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Multimodality high-resolution signals from brain-injured patients | at completion of the study up to 3 years
  The investigators aim to collect multimodality high-resolution physiological signals from brain-injured patients. This is not a hypothesis-driven study but rather a signal database development project with a goal to collect multimodality brain monitoring data to support development and validation of algorithms that will be useful for future brain monitoring devices.

CONTACTS AND LOCATIONS:
Overall Officials: Xiao Hu, Principal Investigator — Emory University
Locations (3):
- United States (3):
  - UC Davis, Davis, California
  - University of California San Francisco, San Francisco, California
  - Emory University, Atlanta, Georgia

IPD SHARING:
Plan to Share IPD: No

DOCUMENTS (1):
  • Informed Consent Form (2025-01-03): https://cdn.clinicaltrials.gov/large-docs/96/NCT04548596/ICF_000.pdf